CLINICAL TRIAL: NCT05301504
Title: A Phase Ib Study to Determine the Safety and Immunogenicity of a Bivalent ChAdOx1 Vectored Vaccine Against Zaire and Sudan Ebola Virus Species in Tanzanian Healthy Adult Volunteers
Brief Title: A Study in Tanzania of a New Vaccine Against Two Types of Ebola
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: EBL08
Record Dates: First submitted 2022-02-24; First posted 2022-03-29 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-11

CONDITIONS: Ebola
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): n=6 participants vaccinated with a single dose of ChAdOx1 biEBOV 5×10^9 vp
  Interventions: Biological: ChAdOx1 biEBOV
- Group 2 (Experimental): n=6 participants vaccinated with a single dose of ChAdOx1 biEBOV 2.5×10^10 vp
  Note: The DSMB may recommend increasing the size of group 2 to n=9 in the event of higher than expected reactogenicity
  Interventions: Biological: ChAdOx1 biEBOV
- Group 3 (Experimental): n=11 participants vaccinated with a single dose of ChAdOx1 biEBOV 5×10^10 vp
  Interventions: Biological: ChAdOx1 biEBOV
- Group 4 (Experimental): n=25 participants vaccinated with a two doses of ChAdOx1 biEBOV at the final selected dose, based on safety data for groups1-3. The second dose is administered after 12 weeks.
  Note:The dose for group 4 will be selected following a review of safety data to 28 days post vaccination for all previous participants (groups 1 to 3
  Interventions: Biological: ChAdOx1 biEBOV

INTERVENTIONS:
Biological: ChAdOx1 biEBOV — ChAdOx1 biEBOV is provided as a liquid in glass vials and administered intramuscularly into the deltoid of the non-dominant arm (preferably)

SUMMARY:
An open label, first in human, non-randomised, dose escalation, single centre, phase Ib clinical trial

DETAILED DESCRIPTION:
This is an open label, first in human, dose escalation, phase Ib clinical trial to assess the safety and immunogenicity of the candidate ChAdOx1 biEBOV vaccine in healthy Tanzanian volunteers aged 18-45. The vaccine will be administered intramuscularly (IM). There will be 4 study groups and it is anticipated that a total of 76 volunteers will be enrolled. Dose escalation and sentinel participant procedures will be implemented. Volunteers will be first recruited into Group 1 and subsequently into Groups 2 and 3 following interim clinical safety reviews. Volunteers will be sequentially allocated to a study group by selecting eligible volunteers for enrolment following screening. Sequential allocation will occur based on the order in which volunteers are enrolled. Group 4 will be recruited last, with dose selection being dependent on completion of groups 1-3 and a review of safety data.

The trial is funded by Innovate UK project reference 971615.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 18 to 45 years.
2. Able and willing (in the Investigator's opinion) to comply with all study requirements.
3. Agreement to release medical and other information concerning contra-indications for participation in the study, and to be attended by a study clinician for physical examination and any other clinical investigations.
4. Agreement to refrain from blood donation while in the study.
5. Able to read and write
6. Provide written informed consent.
7. For women of childbearing potential only: Willingness to practice continuous effective contraception for the duration of the trial
8. For women of childbearing potential only: A negative pregnancy test on the day of both screening and vaccination.
9. Long term (at least 6 months) or permanent residence in Bagamoyo district.
10. Availability through mobile phone 24 hours a day during the whole study period
11. Agreement to provide personal contact information and contact information of a third party
12. household member or close friend to study team.

Exclusion Criteria:

1. Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment or during the trial follow up period.
2. Receipt of a recombinant simian adenoviral vaccine prior to enrolment
3. Planned receipt of another adenoviral vectored vaccine (e.g., Oxford/AstraZeneca or Janssen COVID-19 vaccines) within 90 days after the vaccination with the ChAdOx1 biEBOV
4. Planned or actual receipt of any vaccines administered within 30 days (before or after) enrolment and/or planned receipt of a vaccine ≤30 days after enrolment EXCEPT for protein, RNA (or other non-adenovirus based) COVID-19 vaccinations which may be given within 14 days of the trial vaccine.
5. Previous receipt of an Ebolavirus vaccine
6. Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate.
7. Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) systemically active immunosuppressant medication within the past 6 months.
8. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
9. History of hereditary angioedema acquired angioedema, or idiopathic angioedema.
10. History of anaphylaxis in relation to vaccination.
11. History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
12. History of serious psychiatric condition likely to affect participation in the study.
13. Ongoing or planned pregnancy or breastfeeding during the trial follow up period
14. Known history of bleeding disorder (e.g., Factor deficiency, coagulopathy, or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture.
15. History of confirmed major thrombotic event (including cerebral venous sinus thrombosis, deep vein thrombosis, pulmonary embolism), known history of antiphospholipid syndrome, or history of heparin induced thrombocytopenia.
16. Any other serious chronic illness requiring hospital specialist supervision.
17. Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week.
18. Suspected or known injecting drug abuse in the 5 years preceding enrolment.
19. Detectable circulating hepatitis B surface antigen (HBsAg).
20. Seropositive for hepatitis C virus (antibodies to HCV).
21. Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis.
22. Body mass index (BMI) of <18 or >30 Kg/m2
23. Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.
24. Acute disease at the time of administration of the IMP (acute disease is defined as the presence of a moderate or severe illness with or without fever). All vaccines can be administered to persons with a minor illness such as diarrhoea or mild upper respiratory infection without fever, i.e., axillary temperature < 37.5°C.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Investigate the safety and tolerability of ChAdOx1 biEBOV in healthy volunteers. | 7 days following vaccination
  Occurrence of solicited local reactogenicity signs and symptoms
Investigate the safety and tolerability of ChAdOx1 biEBOV in healthy volunteers. | 7 days following vaccination
  Occurrence of solicited systemic reactogenicity signs and symptoms
Investigate the safety and tolerability of ChAdOx1 biEBOV in healthy volunteers. | 28 days following vaccination
  Occurrence of unsolicited adverse events (AEs)
Investigate the safety and tolerability of ChAdOx1 biEBOV in healthy volunteers. | Days 0, 2, 7, 28
  Occurrence of changes from baseline for safety laboratory measures
Investigate the safety and tolerability of ChAdOx1 biEBOV in healthy volunteers. | Whole duration of the study (~6 months)
  Occurrence of SAEs and AESIs

SECONDARY OUTCOMES:
Investigate the immunogenicity of ChAdOx1 biEBOV in healthy adult volunteers. | Days 0, 28, 56, 182
  Filovirus GP specific serological response as measured by ELISA
Investigate the immunogenicity of ChAdOx1 biEBOV in healthy adult volunteers. | Days 0, 7, 14, 28, 56, 128
  Filovirus GP specific T cell response measured by IFN-γ ELISPOT

CONTACTS AND LOCATIONS:
Locations (1):
- Bagamoyo Clinical Trial Facility, Bagamoyo, Tanzania